CLINICAL TRIAL: NCT05034029
Title: Effect of Metformin on Tibiofemoral Cartilage Volume and Knee Symptoms Among Overweighted Knee Osteoarthritis patients-a Randomized Clinical Trial
Brief Title: Effect of Metformin on Patients With Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K-2021-001-02
Record Dates: First submitted 2021-08-25; First posted 2021-09-05 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-08

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Experimental): Metformin hydrochloride sustained release tablet will administer orally in escalating doses to reduce side-effects and maintain masking: 0.5 g/day for the first two weeks, 1 g/day for the next 2 weeks, and then 2 g/day until the end of the study if tolerated. If the subject cannot tolerate the maximum dose (2 g/day), take their maximum tolerable dose. In case of adverse reaction, the researchers can determine whether the subject needs to reduce or stop the drug based on their discretion.
  Interventions: Drug: Metformin hydrochloride sustained release tablets
- Placebo (Placebo Comparator): Placebo will administer the same as the experimental drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin hydrochloride sustained release tablets — Oral
  Arms: Metformin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This randomized controlled trial aims to investigate if metformin has osteoarthritis protective effects among overweighted knee osteoarthritis patients. The co-primary outcomes are changes in tibiofemoral cartilage volume and Western Ontario and McMaster Universities Arthritis Index (WOMAC) from baseline to month 24. The secondary outcomes are changes in visual analog scale (VAS)-assessed knee pain, tibiofemoral cartilage defect, effusion-synovitis volume, and tibiofemoral bone marrow lesion maximum size from baseline to month 24.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the American College of Rheumatology (ACR) criteria for symptomatic knee osteoarthritis assessed by a rheumatologist;
2. Age 50 to 75 years;
3. Body mass index ≥ 24 kg/m2;
4. Knee pain ≥ 20 on a 100 mm visual analogue scale (VAS);
5. Able to listen, speak, read and understand Chinese; capable of understanding the study requirements and willing to cooperate with the study instructions; able to provide written, informed consent.

Exclusion Criteria:

1. Severe radiographic knee OA as grade 3 joint space narrowing according to the Osteoarthritis Research Society International (OARSI) atlas;
2. Severe knee pain as knee pain ≥ 80 on a 100 mm VAS;
3. Planned knee or hip surgery (including arthroscopy, joint replacement, and joint open operation) within 2 years;
4. Severe knee trauma history (including arthroscopy, severe injury of knee ligament or meniscus);
5. Contraindication to MRI scanning (e.g. implanted pacemaker, artificial metal valve or cornea, aneurysm clipping surgery, arterial dissection, metal foreign bodies in the eyeball, claustrophobia);
6. Other forms of inflammatory arthritis (e.g. rheumatoid arthritis, psoriatic arthritis);
7. Active malignant cancer or other life-threatening diseases;
8. Type 1 or type 2 diabetes mellitus;
9. Clinical manifestation of liver dysfunction or alanine aminotransferase/aspartate aminotransferase exceeding 2 times the upper limit of normal value;
10. Estimated glomerular filtration rate less than 60 ml/min/1.73 m2;
11. Hypoxic state (e.g. chronic heart insufficiency, acute myocardial infarction, heart failure, chronic obstructive pulmonary disease, cor pulmonale, peripheral vascular disease);
12. Alcoholism;
13. Pregnancy or lactation;
14. Allergic to metformin hydrochloride;
15. Conditions affecting the absorption of oral drugs (e.g. postgastrectomy and malabsorption syndrome);
16. Use of metformin in recent 30 days or plan to use metformin in the next 2 years;
17. Use of investigational drug in recent 30 days.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of tibiofemoral cartilage volume from baseline to 24 months follow up | Baseline and 24 months follow up
  Cartilage volume will be automatically calculated based on a standardized view of 3D cartilage geometry by OsiriX software (University of Geneva, Geneva, Switzerland). The 3D cartilage geometry is composed from the 2D cartilage shapes, which are generated by drawing contours around the cartilage boundaries on section-by-section MR images. Tibiofemoral cartilage volume will be calculated as the sum of both the tibial and femoral compartments.
Change of Western Ontario and McMaster Universities Osteoarthritis Index from baseline to 24 months follow up | Baseline and 3, 6, 12, 24 months follow up
  The WOMAC system in a 100-mm visual analog format will be used to quantify the degree of knee pain (5 questions), joint stiffness (2 questions), and physical dysfunction (17 questions) during the last 7 days. The WOMAC score will be calculated by summing the score of each question (1 point for every 1 mm), and a higher score of WOMAC represents a severe OA symptom. The WOMAC score will be considered invalid and treated as missing data if more than 5 of the questions are not answered. In case no more than 5 items are missed, the remaining items will be averaged and then multiplied by 24 to create the WOMAC score.

SECONDARY OUTCOMES:
Change of knee pain visual analog scale from baseline to 24 months follow up | Baseline and 3, 6, 12, 24 months follow up
  The 100 mm VAS will be used to assess the knee pain during the last 7 days, and a higher VAS indicates a severe knee pain.
Change of tibiofemoral cartilage defect from baseline to 24 months follow up | Baseline and 24 months follow up
  Cartilage defects will be graded using a modified Outerbridge classification as follows: grade 0, normal cartilage; grade 1, focal blistering and intra-cartilaginous hyperintensity with a normal contour; grade 2, irregularities on the surface and loss of thickness of less than 50%; grade 3, deep ulceration with loss of thickness of more than 50% without exposure of subchondral bone; grade 4, full-thickness chondral wear with exposure of subchondral bone. Cartilage defects will be assessed at the medial tibial, medial femoral, lateral tibial, and lateral femoral compartments, and tibiofemoral cartilage defects will be obtained by summing the scores of the four compartments.
Change of effusion-synovitis volume from baseline to 24 months follow up | Baseline and 24 months follow up
  Effusion-synovitis volume will be measured at suprapatellar pouch, central portion, posterior femoral recess, and subpopliteal recess according to the anatomy of the knee joint synovial cavity. Effusion synovitis will be isolated by selecting a region of interest with an intra-articular fluid-equivalent signal on the section-by-section 2D MR images. The volume of effusion-synovitis will be generated using OsiriX software. Total effusion-synovitis volume of the knee will be obtained by summing the volume of possible effusion synovitis in the four synovial cavities.
Change of tibiofemoral bone marrow lesion maximum size from baseline to 24 months follow up | Baseline and 24 months follow up
  Bone marrow lesions is defined as discrete areas of increased signal in the subchondral bone. Bone marrow lesions maximum size will be assessed at the medial tibial, medial femoral, lateral tibial, and lateral femoral compartments. Slice with the greatest area of bone marrow lesions in a specific compartment will be chosen to assess bone marrow lesions maximum size of the corresponding compartment. Bone marrow lesions on adjacent slices will be measured and compared to locate the slice with the maximum lesion size. Tibiofemoral bone marrow lesions maximum size will be calculated by summing the maximum lesions size of the four compartments.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Foshan First People's Hospital, Foshan, Guangzhou
  - Guangzhou First People's Hospital, Guangzhou
  - Liwan Central Hospital of Guangzhou, Guangzhou
  - Sun Yat-Sen Memorial Hospital, Guangzhou
  - Zhujiang Hospital, Guangzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruan G, Yuan S, Lou A, Mo Y, Qu Y, Guo D, Guan S, Zhang Y, Lan X, Luo J, Mei Y, Zhang H, Wu W, Dai L, Yu Q, Cai X, Ding C. Can metformin relieve tibiofemoral cartilage volume loss and knee symptoms in overweight knee osteoarthritis patients? Study protocol for a randomized, double-blind, and placebo-controlled trial. BMC Musculoskelet Disord. 2022 May 21;23(1):486. doi: 10.1186/s12891-022-05434-2. PMID 35598008